CLINICAL TRIAL: NCT03127553
Title: Technological and Clinical Innovative Protocols for the Production of Functional Foods - 6.7 (ProAliFun67)
Brief Title: ProAliFun_6.7_Health Effects of a Low-Salt Bread on Hypertensive Subjects (ProAliFun67)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Ospedali Riuniti di Foggia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProAliFun_6.7_CE4373
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
Keywords: salt intake; functional food; low-salt bread; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A - control (No Intervention): Free diet with standard bread
- B - low-salt diet with normal bread (Active Comparator): Low-sodium diet with standard bread
  Interventions: Dietary Supplement: Low-sodium diet with standard bread
- C - low-salt diet with low-salt bread (Experimental): Low-sodium diet with low-sodium bread
  Interventions: Dietary Supplement: Low-sodium diet with low-sodium bread

INTERVENTIONS:
Dietary Supplement: Low-sodium diet with standard bread — low-sodium diet (2300 mg Na/die) with use of standard bread (750 mg Na/100g) for 6 months
  Arms: B - low-salt diet with normal bread
Dietary Supplement: Low-sodium diet with low-sodium bread — low-sodium diet (2300 mg Na/die) with use of low-salt bread (280 mg Na/100g) for 6 months
  Arms: C - low-salt diet with low-salt bread

SUMMARY:
The purpose of this clinical study is to evaluate the health properties of a dietary intervention carried on with an innovative low-salt bread.

The hypothesis is that the introduction of a low-sodium bread as part of a low-salt diet may improve the compliance to the own regime and that the vascular function, the inflammatory and oxidative state, the composition of the intestinal microbiota and that neurocognitive and neurodegenerative processes can improve in hypertensive patients fed a low-salt diet with low-salt bread.

DETAILED DESCRIPTION:
This clinical trial is a multi-center, randomized, controlled, open label, pilot study, lasting 6 months.

A target number of seventy individuals with hypertension meeting inclusion and exclusion criteria, assessed at enrollment, and which have signed the informed consent, will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* arterial hypertension stage I-II
* stable control of blood pressure
* eGFR > 60
* informed consent signed

Exclusion Criteria:

* uncontrolled hypertension
* therapy with diuretics
* need for therapy with more than three antihypertensive drugs
* proteinuria greater than 1 g/day
* celiac disease
* systemic inflammatory diseases
* suspicion or clinical diagnosis of malignancy
* chronic liver disease
* treatment with corticosteroids or immunosuppressive drugs
* previous acute cardiovascular diseases (myocardial infarction, stroke)
* psychiatric conditions reducing the compliance to treatment protocols

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sodium intake | 6 months
  Reduction of sodium intake in diet with the introduction of the innovative formulation of low-salt bread

SECONDARY OUTCOMES:
Blood pressure | 6 months
  Reduction of blood pressure
Endothelial stress | 6 months
  Improvement of flow-mediated dilation FMD
Gut microbiota | 6 months
  Evaluation of gut microbiota modulation
Antioxidant status | 6 months
  Evaluation of the antioxidant/oxidant ratio of blood
Inflammation | 6 months
  State of sub-clinical inflammation
Insulin sensitivity | 6 months
  Reduction of insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, MD Full Prof, Principal Investigator — Head of the Nephrology, Dialysis and Transplantation Unit "Aldo Moro" University of Bari Azienda Ospedaliero-Universitaria Consorziale "Policlinico"
Locations (1):
- AUO Policlinico Consorziale, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosola C, Pesce F, De Angelis M, Maranzano V, Zito A, Montemurno E, Dalfino G, Loiudice S, Creanza V, Pompa G, Ciccone MM, Grandaliano G, Stallone G, Gesualdo L. Effects of low-sodium bread on dietary compliance and fecal cultivable bacteria in a randomized controlled pilot trial in hypertensive subjects. BMC Nutr. 2024 Feb 21;10(1):31. doi: 10.1186/s40795-024-00838-w. PMID 38383476